CLINICAL TRIAL: NCT02495662
Title: The LIPMAT Study: Liposomal Prednisolone to Improve Hemodialysis Fistula Maturation
Acronym: LIPMAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow inclusion
Sponsor: Leiden University Medical Center (Other)
Collaborators: HagaZiekenhuis (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); OLVG (Network); Medical Center Haaglanden (Other); Reinier de Graaf Groep (Other); Spaarne Gasthuis (Other); Alrijne Hospital (Other); Tergooi Ziekenhuis (Unknown)
Responsible Party: Principal Investigator, JorisRotmans, J.I. Rotmans, MD, PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIPMAT
Record Dates: First submitted 2015-07-02; First posted 2015-07-13 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-05

CONDITIONS: Renal Dialysis; Hemodynamics; Vascular Remodeling; Neointima
Keywords: Vascular access; Hemodialysis; Arteriovenous shunt; Arteriovenous fistula; Maturation; Liposomal prednisolone; PEG-liposomal prednisolone sodium phosphate; Radio-cephalic; Shunt
MeSH Terms: conditions — Vascular Remodeling; Neointima; Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposomal prednisolone (Experimental): Treatment with polyethylene glycol (PEG)-liposomal prednisolone sodium phosphate 150mg in 500ml saline intravenously at 1 and 15 days post surgery.
  Interventions: Drug: PEG-liposomal prednisolone sodium phosphate
- Placebo (Placebo Comparator): Treatment with 500ml normal 0.9% saline intravenously at 1 and 15 days post surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PEG-liposomal prednisolone sodium phosphate — Liposomal prednisolone
  Other Names: Nanocort
  Arms: Liposomal prednisolone
Drug: Placebo — 0.9% normal saline
  Arms: Placebo

SUMMARY:
This study will investigate if liposomal prednisolone is effective in promoting arteriovenous fistula (AVF) maturation when administered to human subjects after surgical creation of a radio-cephalic AVF.

DETAILED DESCRIPTION:
AVFs are the preferred means of vascular access for maintenance hemodialysis. Nonmaturation occurs in 30-50% of cases, with highest rates in radio-cephalic fistulas. Inflammatory cytokines are involved in this process of nonmaturation. By suppressing inflammation, corticosteroids might promote maturation, but have significant systemic side effects. Liposomal prednisolone has a long circulation time and targets inflamed tissue with low systemic concentrations and limited side effects. In an animal study, it was demonstrated to promote AVF maturation. At present, no drug therapy aimed at improving shunt maturation is available. This study will investigate if liposomal prednisolone is effective in promoting AVF maturation when administered to human subjects after surgical creation of a radio-cephalic AVF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are scheduled for creation of a radiocephalic AVF for maintenance hemodialysis.
2. Male or female ≥ 18 years old.
3. Patients are able and willing to give written informed consent.

Exclusion Criteria:

1. Any concurrent illness, disability or clinically significant abnormality that may, as judged by the investigator, affect the interpretation of clinical efficacy or safety data or prevent the subject from safely completing the assessments required by the protocol.
2. Current participation in another interventional clinical trial or subjects who have received an investigational drug within 30 days prior to the baseline visit.
3. History of psychosis.
4. History of osteonecrosis
5. Previous AVF in the ipsilateral arm.
6. Current central venous catheter at the ipsilateral side.
7. Treatment with oral, rectal or injectable (including intra-articular) glucocorticoids (CS) within 6 weeks prior to baseline visit. Inhaled glucocorticoids are allowed. Topical steroids are allowed, however subjects should not have received more than 100 gram of a mild to moderate topical corticosteroid cream per week, 50 gram of a potent corticosteroid cream per week or 30 gram of a very potent topical corticosteroid cream per week in the 4 weeks prior to the baseline visit.
8. Treatment with immunosuppressant drugs. Treatment with non-steroidal anti-inflammatory drugs (NSAIDs).
9. Patients who are unlikely to adequately comply with the trial's procedures (due for instance to medical conditions likely to require an extended interruption or discontinuation, history of substance abuse or noncompliance).
10. Women who are lactating, pregnant (positive pregnancy test at baseline) or planning to become pregnant during the course of the study.
11. Unwillingness to use reliable and acceptable contraceptive methods throughout the study and till 3 months after last study medication except for female patients who are surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) or at least 1 year postmenopausal.
12. Malignant disease, unless cured. Current prostate carcinoma without current or planned cytostatic therapy is allowed.
13. Uncontrolled Diabetes mellitus.
14. Signs of active infection, requiring systemic treatment.
15. Positive Quantiferon test.
16. Subject with positive hepatitis panel (including hepatitis B surface antigen [HBsAg], and / or anti-hepatitis B core antibodies, and / or hepatitis C virus antibody [anti-HCV]).
17. History of anaphylaxis or severe allergic responses, including to radio-contrast agents.
18. Planned live-virus vaccinations.
19. Planned surgical interventions or planned elective hospital admissions within 6 weeks after AVF surgery. Planned hemodialysis sessions do not count as an exclusion criterion.
20. Abnormal hepatic function (Alanine aminotransferase (ALT)/ aspartate aminotransferase (AST) or bilirubin > 2 x upper limit of normal) at the time of the screening visit.
21. Clinically significant out-of-range values on hematology panel, at discretion of the Principal Investigator.
22. Current substance abuse or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Cephalic vein diameter | 6 weeks after surgical creation of the radiocephalic shunt.
  Echographic measurement of the diameter of the cephalic vein, six weeks after surgical creation of the radiocephalic shunt.

SECONDARY OUTCOMES:
Cephalic vein diameter | 3 months after surgical creation of the radiocephalic shunt.
  Echographic measurement of the diameter of the cephalic vein, three months after surgical creation of the radiocephalic shunt.
Radial artery diameter | 6 weeks after surgical creation of the radiocephalic shunt.
  Echographic measurement of the diameter of the radial artery, six weeks after surgical creation of the radiocephalic shunt.
Radial artery diameter | 3 months after surgical creation of the radiocephalic shunt.
  Echographic measurement of the diameter of the radial artery, three months after surgical creation of the radiocephalic shunt.
Radial artery flow. | 6 weeks after surgical creation of the radiocephalic shunt.
  Echographic measurement of the flow of the radial artery, six weeks after surgical creation of the radiocephalic shunt.
Radial artery flow. | 3 months after surgical creation of the radiocephalic shunt.
  Echographic measurement of the flow of the radial artery, three months after surgical creation of the radiocephalic shunt.

CONTACTS AND LOCATIONS:
Overall Officials: Joris I Rotmans, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No